CLINICAL TRIAL: NCT03165201
Title: Non-invasive Rapid Assessment of Patients With Liver Transplants Using Magnetic Resonance Imaging With LiverMultiScan.
Acronym: RADIcAL2
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Collaborators: Leiden University Medical Center (Other); University of Coimbra (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PJM126
Record Dates: First submitted 2017-05-18; First posted 2017-05-24 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation and Biopsy; Liver transplantation and LiverMultiScan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional serum biobanking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LiverMultiScan — We will study participants who are due to be evaluated for possible liver transplant rejection. There will be no change to usual care as part of the study, but patients will get an additional MRI scan, so that the results can be compared to the biopsy results. Each centre has a consultant radiologist specialising in liver imaging with experience in post-transplant review; the radiologist will review the MRI scans and inform the patient's doctor if any structural liver abnormalities are found (e.g. abnormal vessels, haemangiomas, tumours or cysts) as this may have implications for the patient's planned biopsy.

SUMMARY:
This will be a prospective, multi-centre, biomarker trial comparing the accuracy of a new test (LiverMultiScan) against an existing test (liver biopsy) in the assessment of liver transplant recipients, designed in accordance with the STARD criteria.

Study participants are 200 patients with liver transplant, due to undergo liver biopsy as part of serial evaluation of their liver health and to rule out rejection. The whole study will take 3 years with 2 years of recruitment The main aim is to investigate whether the introduction of LiverMultiScan as a standardised diagnostic test for liver disease can match the diagnostic yield of existing biopsies.

DETAILED DESCRIPTION:
Long-term survival after solid organ transplantation has increased during the last decade due to improvements in surgical technique, peri-operative care, and more efficient immunosuppression (IS) (1). However, transplant recipients still exhibit higher morbidity and mortality than the general population. One of the main causes are co-morbidities which are negatively influenced by chronic IS drug usage. It is however a very fine balance, as under-usage of IS can lead to transplant rejection (2). Therefore, many paediatric and some adult liver transplant recipients have regular liver biopsies as part of their serial evaluation, so-called 'routine liver biopsies'. Biopsy is performed if there is suspected rejection, as no current non-invasive tests are both sensitive and specific for rejection. Biopsy is used to identify early histological signs of rejection. However, there are some problems;

* There is a risk of complication due to biopsy(1 in 10,000)
* biopsies are painful
* sample only a tiny fraction of the liver and for children there is a need to sedate.

Therefore, they are less-than-perfect for serial evaluation. Optimisation of IS has become a priority goal in transplantation, but is hampered by the lack of diagnostic tests available for serial monitoring (3). There are potential benefits of IS minimization or withdrawal, however this need to be balanced with the risks, inconveniences and costs of prompting liver allograft rejection.

Identification of a reproducible and reliable non-invasive assessment tool for the transplanted liver, such as multiparametric quantitative MRI, would therefore substantially benefit the liver transplant population. In Europe, approximately 6000 liver transplants are performed every year (1). Under the current standard-of-care, indefinite pharmacological IS is prescribed to all of them. The cost of immunosuppressive drugs is €4200- €7000 per patient per year (£3000-£5000/patient/year). In addition to its cost, chronic IS may result in substantial side effects (hypertension, diabetes, renal insufficiency, hyperlipidaemia, cancer, infections) that contribute to patient morbidity and mortality (2). Rejection is a major concern with liver transplant recipients. At present, there is no clear non-invasive diagnostic pathway to identify early rejection. We would like to see if the implementation of LiverMultiScan (4) to monitor the transplant population and modify treatment can replace or equal the yield of invasive liver biopsies in the post-transplant population.

Therefore, the aim of this study is to determine whether there is concordance between using LiverMultiScan and liver biopsy in a post-liver transplant population.

The primary objective is to investigate whether the introduction of LiverMultiScan as a standardised diagnostic test for liver disease can match the diagnostic yield of existing biopsies.

The following are the secondary objectives;

* To determine patient feedback from this population (transplant recipients) on LiverMultiScan.
* To assess how multiparametric MRI correlates with other measures of fibrosis and rejection (eg elastography, blood tests) in the evaluation of these patients.
* To evaluate the utility of LMS in the diagnosis of de novo or recurrent liver disease post transplant
* To evaluate biliary changes in post-transplant patients with quantitative MRCP

Patients who meet the inclusion criteria will be approached by a member of their clinical care team and asked if they are interested in taking part in the study. Both adult and paediatric patients with a liver transplant due to have a liver biopsy, being seen in medical/gastroenterology clinic, will be invited to take part in the study.

Once a potential adult participant has expressed interest in the study, he/she will be provided with a PIL (Patient Information Leaflet) and an opportunity to discuss his/her eligibility and the details of the study with her family and doctor.

Age-appropriate written and verbal versions of the PIL and Informed Consent will be presented to the paediatric participants and their guardians. Once the participants and/or their guardians (as appropriate) have had time to consider the PIL (minimum 24 hr) and the opportunity to discuss the study with their family, friends and GP, they will be contacted by a member of the study team to check whether they would like to take part and to schedule a study visit. At this point, the inclusion criteria will be explained to all potential female participants of childbearing potential age, that they will not be able to take part in the study if they are pregnant.

The informed consent process will be carried out during the first study visit.

Informed consent to have an extra MR scan in addition to usual care will be sought by an appropriately trained member of the study team. Age-appropriate written and verbal versions of the Participant Information and Informed Consent presented to the participants and their guardians detailing no less than:

* The exact nature of the study;
* what it will involve for the participant;
* the implications and constraints of the protocol;
* and any risks involved in taking part.

It will be clearly stated that the participant is free to withdraw from the study at any time for any reason without prejudice to future care, and with no obligation to give any reason for withdrawal.

The participant will be allowed as much time as they wished to consider the information, and the opportunity to ask questions from the Investigator, their GP or other independent parties to decide whether they will participate in the study. Written Informed Consent will then be obtained by means of participant-dated signature and dated signature of the person who presented and obtained the Informed Consent. In the case of minors under 16 years of age, consent will be taken from at least one guardian and assent from the child age 6 and above. For adolescents aged 16-18, consent will be taken from the adolescents themselves. GPs will also be informed about patient taking part in the study, with participants' consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 6 yrs old with a liver transplant.
* Patients due to undergo routine liver biopsy or biopsy for suspected pathology after liver transplantation
* Patients (and / or Guardians) who are willing and able to give informed consent for participation in the study.

Exclusion Criteria:

The participant may not enter the study if they have any contraindication to magnetic resonance imaging (inc pregnancy, pacemaker, shrapnel injury, severe claustrophobia). We will record the number of patients who have to be excluded for those reasons (expected to be <5%).

Children / adults with a contraindication to liver biopsy (coagulopathy, obstructed biliary tract with high risk of bile leak, ascites etc).

Children or adults who are unable to tolerate MRI without sedation or general anaesthetic.

Ages: 6 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 150 adults, and 50 children and adolescents with liver transplant, who are due to undergo liver biopsy as part of serial evaluation of their liver health or for suspected pathology.
  Patients who meet the inclusion criteria will be approached by a member of their clinical care team and asked if they are interested in taking part in the study. Both adult and paediatric patients with a liver transplant due to have a liver biopsy, being seen in medical/gastroenterology clinic, will be invited to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
The cT1 (inflammation) measured by LMS compared to biopsy results, to assess fibro-inflammatory status and rejection status | 12 months
  To investigate whether the introduction of LiverMultiScan as a standardised diagnostic test for liver disease can match the diagnostic yield of existing biopsies.

SECONDARY OUTCOMES:
Patient feedback on LiverMultiScan | 1 Year
  To determine patient feedback from this population (transplant recipients) on LiverMultiScan.
Correlation of diagnostic tests. | 1 Year
  To assess how multiparametric MRI correlates with other measures of fibrosis and rejection (eg. elastography, blood tests) in the evolution of these patients.
LiverMultiScan utility | 1 year
  To evaluate the utility of LMS in the diagnosis of de novo or recurrent liver disease post transplant.
Biliary changes using MRCP. | 1 Year
  To evaluate biliary changes in post-transplant patients with quantitative MRCP.

CONTACTS AND LOCATIONS:
Overall Officials: Minneke Coenraad, MD, Principal Investigator — Leiden University Medical Centre; Emer Fitzpatrick, MD, Principal Investigator — King's College Hospital NHS Trust
Locations (3):
- Leiden University Medical Center, Leiden, South Holland, Netherlands
- University of Coimbra, Coimbra, Centro, Portugal
- King's College Hospital, London, Brixton, United Kingdom

IPD SHARING:
Plan to Share IPD: No